CLINICAL TRIAL: NCT02753712
Title: A Two-arm, Randomised, Assessor-blind, Parallel Group Study to Evaluate the Effect of Fluticasone/Formoterol Breath Actuated Inhaler (BAI) and Relvar® Ellipta® DPI on Ventilation Heterogeneity in Subjects With Partially Controlled or Uncontrolled Asthma
Brief Title: A Study to Evaluate the Effect of Fluticasone/Formoterol Breath Actuated Inhaler (BAI) or Relvar® Ellipta® DPI on Ventilation Heterogeneity in Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFL3502; 2015-000801-38 (EudraCT Number)
Record Dates: First submitted 2016-04-11; First posted 2016-04-28 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Asthma
Keywords: Small airway disease; asthma
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fluticasone/vilanterol DPI (Relvar Ellipta DPI) (Active Comparator): Inhalation powder. 92/22µg, I inhalation od
  Interventions: Drug: Fluticasone/Vilanterol DPI (Relvar Ellipta DPI)
- Fluticasone/formoterol BAI (Experimental): Pressurised suspension for inhalation 125/5µg, 2 inhalations bid
  Interventions: Drug: Fluticasone/Formoterol BAI

INTERVENTIONS:
Drug: Fluticasone/Formoterol BAI
  Arms: Fluticasone/formoterol BAI
Drug: Fluticasone/Vilanterol DPI (Relvar Ellipta DPI)
  Arms: fluticasone/vilanterol DPI (Relvar Ellipta DPI)

SUMMARY:
The purpose of this study is to demonstrate improvement of peripheral airway resistance (R5-R20) from baseline with fluticasone/formoterol breath actuated inhaler (BAI).

ELIGIBILITY:
Inclusion Criteria for subjects on Seretide Accuhaler 250/50 µg at screening:

1. Male and female subjects ≥18 years old.
2. Adequate contraception
3. Documented clinical history of asthma for ≥6 months prior to screening visit
4. Using Seretide Accuhaler at a stable dose of 250/50 μg BID at screening for ≥ 8 weeks.
5. uncontrolled asthma as defined by Asthma Control Questionnaire (ACQ-6) score ≥ 1.0
6. R5-R20 ≥ 0.10 kPa/L/s as measured on impulse oscillometry during the screening visit.
7. Historical evidence (within 24 months) of eosinophilic airways disease evidenced by sputum eosinophil count ≥ 3% and/or FeNO 35 ppb.

Inclusion criteria for subjects on equivalent /higher dose or other ICS-LABAs or higher dose of Seretide at screening:

1. Male and female subjects ≥18 years old.
2. Adequate contraception
3. Documented clinical history of asthma for ≥6 months prior to screening visit
4. R5-R20 ≥0.07 kPa/L/s as measured on impulse oscillometry during the screening visit.

   * 5. Historical evidence (within past 24 months) of eosinophilic airways disease, evidenced by sputum eosinophil count ≥3% and/or FeNo ≥35 ppb.

Exclusion Criteria for all subjects:

1. Any severe chronic respiratory disease other than asthma.
2. Subject has a smoking history ≥10 "pack years" (i.e., at least 1 pack of 20 cigarettes/day for 10 years or 10 packs/day for 1 year, etc.)
3. Current smoking history within 12 months prior to the screening visit
4. Near fatal or life-threatening (including intubation) asthma within the past year.
5. Known history of systemic (injectable or oral) corticosteroid medication within 1 month of visit 1.
6. Evidence of a clinically unstable disease as determined by medical history or physical examination that, in the investigator's opinion, precludes entry into the study. 'Clinically unstable' is defined as any disease that, in the opinion of the Investigator, would put the subject at risk through study participation, or which would affect the outcome of the study.
7. In the investigator's opinion a clinically significant upper or lower respiratory infection within 4 weeks prior to visit 1.
8. Current evidence or known history of alcohol and/or substance abuse within 12 months prior to the screening visit.
9. Subject has taken β-blocking agents, tricyclic antidepressants, monoamine oxidase inhibitors, astemizole, quinidine type antiarrhythmics, or potent CYP 3A4 inhibitors such as ketoconazole within 1 week prior to screening visit.
10. Current use of bronchodilators / anti-inflammatory agents other than those specified in the protocol.
11. Known or suspected sensitivity to study drug or excipients.
12. Participation in a clinical drug study within 30 days of the screening visit.
13. Current participation in a clinical study.

Exclusion Criteria for subset of subjects undergoing OR-MRI and HD-CT

1. Contraindication for MRI scanning (as assessed by local MRI safety questionnaire), which includes, but is not limited to: presence of non-MRI compatible artificial heart valves, hydrocephalus shunts, intracranial aneurysm clips, joint replacements or metal implants, pacemakers or other cardiac rhythm management devices, claustrophobia, history of metal in the eye, presence of shrapnel from a war injury, callipers or braces, dentures, dental plates or hearing aids that include metal and cannot be removed, history of epilepsy or black-outs, ear implants, piercings cannot be removed, intrauterine contraceptive device or coil.
2. Inability to stay in the supine position for the duration of the scanning procedure
3. Obesity (body weight >140kg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-14 (Actual)

PRIMARY OUTCOMES:
Measuring peripheral airway resistance (R5-R20) | From baseline to week 8
  Measuring peripheral airway resistance (R5-R20)

SECONDARY OUTCOMES:
measure ventilation heterogeneity (using Functional Respiratory Imaging) | From baseline to week 9
  measures of ventilation heterogeneity
Measuring distal airway volume and resistance (using impulse oscillometry) | From baseline to week 8 and 9
  Measuring distal airway volume and resistance (using Functional Respiratory Imaging (FRI)
Evaluate asthma control (using ACQ-6) ) | From baseline to week 4 and 8
  Evaluate asthma control (using ACQ-6) )
Evaluate health status (using AQLQ) | From baseline to week 4 and 8
  Evaluate health status (using AQLQ)

CONTACTS AND LOCATIONS:
Locations (16):
- Australia (3):
  - The Woolcock Institute of Medical Research, Glebe, New South Wales
  - Epworth Eastern Medical Centre, Box Hill, Victoria
  - Allergy immunology and Respiratory medicine, The Alfred Hospital, Melbourne, Victoria
- New Zealand (2):
  - The New Zealand Respiratory and Sleep Institute, Greenlane, Auckland
  - Otago Respiratory Research Unit, Dunedin
- Slovakia (6):
  - INSPIRO, s.r.o. Ambulancia pneumológie a ftizeológie, Humenné
  - DAMIZA, s.r.o. Ambulancia pneumológie a ftizeológie, Námestovo
  - Poliklinika ADUS, Pľúcna ambulancia, Poprad
  - PULMO, s.r.o, Prešov
  - Pľúcna ambulancia Hrebenár, s.r.o., Spišská Nová Ves
  - ANA JJ, s.r.o, Ambulancia klinickej imunológie a alergológie, Topoľčany
- Skane University Hospital, Lund, Sweden
- United Kingdom (4):
  - Respiratory Biomedical Research Unit, Glenfield Hospital, Leicester, Leicestershire
  - Bradford Teaching Hospital, Bradford
  - Royal Brompton and Harefield Foundation Trust, London
  - University Hospital of South Manchester, Manchester

REFERENCES:
- See also: Link to Eu CT Register — https://www.clinicaltrialsregister.eu/ctr-search/search?query=KFL3502